CLINICAL TRIAL: NCT03208530
Title: A Pilot Study to Test the Acceptability and Feasibility of Brief Motivational Interview Intervention to Help Patients Formulate Their Goals for Medical Care in the Emergency Department
Brief Title: Motivational Interview Intervention to Help Patients Formulate Their Goals for Medical Care in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Kei Ouchi, Principal Investigator, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2016P002637
Record Dates: First submitted 2017-07-03; First posted 2017-07-05 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Emergency Service, Hospital; Motivational Interviewing; Advance Care Planning
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): This is a single arm study with all enrolled patients receiving the same brief motivational interview intervention.
  Interventions: Behavioral: Brief motivational interview intervention

INTERVENTIONS:
Behavioral: Brief motivational interview intervention — A brief (<7minutes) interview by an emergency department clinician to empower patients to formulate and communicate their goals for medical care with patients' outpatient clinicians.

SUMMARY:
Test the acceptability and feasibility of a brief motivational interview intervention to facilitate advance care planning (ACP) conversations for older adults with serious co-morbid illness being discharged from the emergency department (ED). The investigators will interview the participants to understand their perception of the intervention and collect patient-reported outcomes data after leaving the ED.

DETAILED DESCRIPTION:
This study is designed to engage seriously ill older adults in conversations about their goals of care. Our intervention is intended to help these patients understand the significance of ED visits in the course of their illnesses.

ELIGIBILITY:
Inclusion Criteria:

* ≥65 years of age
* English-speaking
* Capacity to consent
* AND ≥1 Serious illness (New York Heart Association stage 3 or 4 heart failure, oxygen-dependent chronic obstructive lung disease, chronic kidney disease on dialysis, and metastatic cancer.) OR determined by the emergency department provider that the patient has a high likelihood of death in the next 12 months ("I would not be surprised if this patient died in the next 12 months.").

Exclusion Criteria:

* Acute physical or emotional distress
* Determined by emergency department provider not to be appropriate
* Clearly documented goals for medical care already exists (e.g. medical order for life sustaining treatment - MOLST).
* Already enrolled in this study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kei Ouchi, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Ouchi K, George N, Schuur JD, Aaronson EL, Lindvall C, Bernstein E, Sudore RL, Schonberg MA, Block SD, Tulsky JA. Goals-of-Care Conversations for Older Adults With Serious Illness in the Emergency Department: Challenges and Opportunities. Ann Emerg Med. 2019 Aug;74(2):276-284. doi: 10.1016/j.annemergmed.2019.01.003. Epub 2019 Feb 13. PMID 30770207

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 75
Completed | 48
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 75
Age, Continuous [Mean (Full Range); unit: years] | 72.68 [39 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 60
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 75

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Found the Intervention Acceptable and Provided Suggestions for Improvement
Description: The investigator will measure quantitatively and qualitatively whether patients found this intervention acceptable and provided suggestions for its improvement.
Time Frame: Immediately following the intervention in the emergency department.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 48
Participants | 48

2. Secondary Outcome: Acceptability of the Intervention by Administering Clinicians.
Description: The investigators will ask the emergency department clinicians who administered the intervention to report the intervention acceptability using a Likert scale survey.
Time Frame: Immediately following the intervention in the emergency department.
Population: The clinicians administrating the intervention are part of the research team and are not subjects of the clinical trial per NIH definition because they are not prospectively assigned to an intervention (they are the intervention itself), and the outcomes assessed from them were not health-related. The mean acceptability using a Likert scale (0 not acceptable, 1-4 somewhat unacceptable, 6-9 somewhat acceptable, and 10 completely acceptable).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 14
score on a scale | 7 (1)

3. Secondary Outcome: Patient's Quality of Life
Description: The investigators will measure patient's quality of life using a validated survey measure (Quality of life at the end of life, QUAL-E, Steinhauser et al. 2004) at baseline and after the intervention. QUAL-E consists of 25-items and measures 4 domains (symptom impact, relationship with the healthcare provider, preparation for the end of life, and life completion). Each item is in a 5-point Likert scale ranging from (1 Not at all to 5 Completely), and lower scores indicate better outcomes for all domains except for the preparation for the end of life domain and life completion domain where higher scores indicate better outcomes. The mean composite score is compared between baseline and 1 month after the intervention.
Time Frame: At baseline (in-person) and 1 month after (over the phone) the intervention.
Population: Patients found this survey too long to complete when they just left the emergency department after acute health decline. Further, the questions were making patients think more about the end of life, which may skew our aim. Therefore, we decided to stop collecting this outcome after the first 9 patients. Only 3 out of those 9 participants completed their 1-month QUAL-E assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 9
score on a scale
  Baseline Overall Score (Mean) | 3.69 (0.28)
  1-month Overall Score (Mean): number analyzed (Participants) | 3
  1-month Overall Score (Mean) | 3.72 (0.20)
  Baseline Symptoms Impact Subscale (Mean) | 3.70 (0.14)
  1-month Symptoms Impact Subscale (Mean): number analyzed (Participants) | 3
  1-month Symptoms Impact Subscale (Mean) | 3.00 (0.98)
  Baseline Relationship with Healthcare Provider Subscale (Mean) | 4.00 (0.71)
  1-month Relationship with Healthcare Provider Subscale (Mean): number analyzed (Participants) | 3
  1-month Relationship with Healthcare Provider Subscale (Mean) | 4.40 (0.60)
  Baseline Preparation for the End of Life Subscale (Mean) | 2.60 (0.31)
  1-month Preparation for the End of Life Subscale (Mean): number analyzed (Participants) | 3
  1-month Preparation for the End of Life Subscale (Mean) | 2.58 (0.96)
  Baseline Life Completion Subscale (Mean) | 4.00 (0.33)
  1-month Life Completion Subscale (Mean): number analyzed (Participants) | 3
  1-month Life Completion Subscale (Mean) | 4.14 (0.50)

4. Secondary Outcome: Advance Care Planning Engagement Behavior
Description: The investigators will measure patient's behaviors and actions for completing advance care planning using a validated survey measure (advance care planning engagement survey, Sudore et al 2017) at baseline and after the intervention. The measure is a 4-item survey measuring actions and behaviors of advance care planning. The additive composite score is calculated and ranges from 1 (least engagement) to 5 (most engagement).
Time Frame: At baseline (in-person) and 1 month after (over the phone) the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 51
score on a scale
  Baseline | 3.8 (0.8)
  Post-intervention (3 month) | 4.3 (0.9)

5. Secondary Outcome: Patient Empowerment
Description: The investigators will measure patient empowerment by using a validated survey measure (Patient Activation Measure, PAM™) at baseline and after the intervention.
Time Frame: At baseline (in-person) and 1 month after (over the phone) the intervention.
Population: We did not collect this outcome as the "advance care planning engagement survey" was felt to be better suited for this study.
Arm/Group | Intervention Arm
Number analyzed (Participants) | 0

6. Secondary Outcome: Patient Distress
Description: The investigators will measure patient anxiety/distress regarding a particular event (in this case, our intervention) by using a validated survey measure (Impact of Event Scale - Revised, IES-R, Weiss 1996) within a week after the intervention. IES-R is a 22-item, 5-point Likert scale measure (ranging from 0 Not at all to 4 Extremely).
  Results consist of the mean rating for the total score and raw scores for three subscales:
  The Avoidance Scale, Intrusion Scale, and the Hyperarousal Scale.
  The scores give an indication of the level of impairment from post traumatic stress, where: 0 = No symptoms 1 = Few symptoms 2 = Moderate symptoms 3 = A High level of symptoms 4 = An Extremely high level of symptoms
Time Frame: Within 7 days after the intervention.
Population: We stopped collecting this outcome after the first 8 patients because patients did not express any clinically meaningful anxiety/distress due to our intervention. Furthermore, a much more traumatic event for these patients seemed to be the recent emergency department visit or hospitalization, which made this scale not appliable.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 8
score on a scale
  Total Score | 0.66 (0.63)
  Subscale - Intrusion | 0.70 (0.61)
  Subscale - Avoidance | 0.86 (1.19)
  Subscale - Hyperarousal | 0.33 (0.31)

ADVERSE EVENTS:
Time Frame: AEs were collected up to the 3 months after the intervention.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 5/75
Serious Adverse Events (participants affected / at risk) | 0/75
Other Adverse Events (participants affected / at risk) | 0/75

LIMITATIONS AND CAVEATS:
We did not collect some pre-specified outcomes because initial data suggested that they may not be clinically relevant.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/30/NCT03208530/Prot_SAP_007.pdf
  • Informed Consent Form: Study Information Sheet for Patients (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT03208530/ICF_008.pdf
  • Informed Consent Form: Study Information Sheet for Clinicians (2017-05-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03208530/ICF_009.pdf